CLINICAL TRIAL: NCT04033016
Title: The Influence of Motivational Public Health Intervention for Improvement of Physical Activity During Pregnancy
Brief Title: Use of Motivational Interviewing for Promotion of Physical Activity During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Todorovic Jovana, teaching assistant, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MI and pregnancy PA
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facebook and motivational interviewing group (Experimental): Women from this group were included in social media intervention and in two sessions of motivational interviewing.
  Interventions: Behavioral: motivational interviewing; Behavioral: online social media intervention
- Facebook only group (Experimental): Women from this group were included in the social media intervention only.
  Interventions: Behavioral: online social media intervention
- control group (No Intervention): women from this group only received the information on the benefits of physical activity during pregnancy.

INTERVENTIONS:
Behavioral: motivational interviewing — Motivational interviewing (MI) is a contemporary form of advisory support, which is often used for behavioral change. During the motivational interviewing educated health professional leads the counseling session by asking questions on lifestyle, attitude towards the behavioral change, and factors pro and against the change. During the MI the focus is on the patient/ client, his/her own perception of their health, understanding the reasons for current behavioral patterns, and encouragement to assess these patterns.
  Arms: Facebook and motivational interviewing group
Behavioral: online social media intervention — Facebook group was specially designed for purposes of intervention and was administered by the research team. It was used to motivate the participants to be more physically active. The intervention used hybrid approach, with health promotion campaign with motivational messages and pictures, journal articles, questions with the aim to spark a discussion on barriers or possibilities for physical activity and participatory approach (all members were allowed to post motivational messages or questions for their peers).
  Arms: Facebook and motivational interviewing group; Facebook only group

SUMMARY:
We conducted a randomized control trial to assess the differences in the increase in PA among pregnant women who were included in the online social media intervention (Facebook group), the combination of online social media intervention and MI (Facebook and MI group) and control group. The study was conducted from January 2018 to April 2019 at the Clinic for Gynecology and Obstetrics, Clinical Centre of Serbia and Institute of Social Medicine, Medical Faculty, University of Belgrade. The women were approached after the prenatal screening at the 12th week of gestation. The intervention lasted through the second trimester. The reassessment was done at the end of the second trimester. The final analysis included 134 women.

DETAILED DESCRIPTION:
The study was designed as a randomized controlled clinical trial and was conducted from January of 2018 to April 2019, at the Clinic for Gynaecology and Obstetrics, Clinical Centre of Serbia, Belgrade and the Institute for Social Medicine, Medical Faculty, University of Belgrade. The study compared the physical activity in the second trimester of pregnancy of the pregnant women who were included in the intervention groups (Facebook group and Facebook and MI group) and pregnant women from the control group. The intervention lasted for three months (from 12th till 28th week of gestation).

Total of 227 women were approached after the double test screening at the end of the first trimester (12th week of gestation). All women without medical or obstetric contraindications for physical activity were included in the study.

Baseline questionnaire consisted of 85 questions divided into five sections: social characteristics (age, place of residence, marital status, education, employment status, self-rated health, self-perceived financial status), anthropometric characteristics (height, weight, waist circumference), pregnancy and lifestyle characteristics (planning a pregnancy, symptoms present during the first trimester, and diet), and physical activity (leisure-time physical activity in the period of three months before pregnancy and physical activity during the first trimester).

At the baseline level, participants filled in the questionnaire and anthropometric measures were recorded. Anthropometric measures, height, weight and waist circumference, were measured by one of the researchers. Randomization was done after the initial baseline measurements. The follow-up measurement was done three months after the baseline, and all participants were asked to fill in the questionnaire which referred to physical activity in the second trimester.

The intervention involved social media intervention and Motivational interviewing.

Facebook group was specially designed for purposes of intervention and was administered by the research team. It was used to motivate the participants to be more physically active. The intervention used a hybrid approach. Motivation was done through health promotion campaign with motivational messages and pictures, journal articles, questions with the aim to spark a discussion on barriers or possibilities for physical activity ('What is your favourite form of physical activity?', 'Do you think that physical activity is safe during pregnancy?', 'Would you like to be more active during pregnancy?', etc). Facebook discussion group used a participatory approach and all members were allowed to post motivational messages or questions for their peers. The reports and photos from organized events (walking, yoga) were also posted regularly, so all participants could follow the level of participation of others. The research team shared information on free sports activities for pregnant women in multiple sports centres in Belgrade, as well as, specially organized events (walking around the lake, yoga).

Women who were randomized in the MI group went through two sessions of MI with the principal researcher. The first MI session was scheduled in the week after the inclusion in the study and the second was after 10-14 days. Each session lasted between 30 and 45 minutes. The principal researcher, who conducted the MI went to certified international training in MI.

ELIGIBILITY:
Inclusion Criteria:

* Women without medical or obstetric contraindication for physical activity during pregnancy.

Exclusion Criteria:

* known medical or obstetric contraindication for physical activity during pregnancy;
* heavy smoking (>20 cigarettes per day)
* mental inability to understand and fill in the questionnaire.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Leisure time physical activity in second trimester | 3 months
  leisure time physical activity is expressed in MET-minutes/week, which is a measure of energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Jovana S Todorovic, MD, Principal Investigator — University of Belgrade, Faculty of Medicine, Institute of Social Medicine; Miroslava Gojnic-Dugalic, MD, PhD, Study Chair — Clinical Center of Serbia, Clinic for Gynecology and Obstetrics
Locations (1):
- Clinical Center of Serbia, Clinic for Gynecology and Obstetrics, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided